CLINICAL TRIAL: NCT03406299
Title: Phase II Randomized Trial of S-1, Leucovorin, Oxaliplatin and Gemcitabine (SLOG) vs Gemcitabine and Cisplatin (GC) in Locally Advanced or Metastatic Biliary Tract Cancer
Brief Title: Phase II Randomized Trial of SLOG vs GC in Locally Advanced or Metastatic Biliary Tract Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T3217
Record Dates: First submitted 2018-01-07; First posted 2018-01-23 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-04

CONDITIONS: Biliary Tract Neoplasms
Keywords: SLOG
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Tegafur; S 1 (combination); Leucovorin; Oxaliplatin; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SLOG regimen (Experimental): Arm 1 interventions : SLOG regimen: treatment for every 14 days as one cycle Tegafur (S-1) 35 mg/m2/b.i.d., day 1 - 7 (maximum dose: 120 mg/day) Leucovorin 30 mg/b.i.d., day 1-7; Oxaliplatin 85 mg/m2 in 250 mL of 5% Glucose, given as 2-hour intra- venous infusion, day 1; Gemcitabine 800 mg/m2 in 250 mL of normal saline, given as fixed dose-rate (FDR, 10 mg/m2/min) infusion, day 1; After the administration of gemcitabine, the infusion line should be flushed with 20 ml of normal saline and then 50 ml of 5% glucose solution before the administration of oxaliplatin
  Interventions: Drug: Tegafur; Drug: Leucovorin; Drug: Oxaliplatin; Drug: Gemcitabine
- GC regimen (Active Comparator): Arm 2 interventions : GC regimen: treatment for every 21 days as one cycle Gemcitabine 1000 mg/m2 in 100 mL of normal saline, IV drip for 30 mins on D1 and D8 Cisplatin 25 mg/m2 in 250ml of normal saline, IV drip for 2 hours on D1 and D8
  Interventions: Drug: Cisplatin

INTERVENTIONS:
Drug: Tegafur — Tegafur(S-1) 35 mg/m2/b.i.d., day 1 - 7 (maximum dose: 120 mg/day)
  Other Names: S-1
  Arms: SLOG regimen
Drug: Leucovorin — Leucovorin 30 mg/b.i.d., day 1-7
  Other Names: Folinic acid
  Arms: SLOG regimen
Drug: Oxaliplatin — Oxaliplatin 85 mg/m2 in 250 mL of 5% Glucose, given as 2-hour intra- venous infusion, day 1
  Other Names: oxalic
  Arms: SLOG regimen
Drug: Gemcitabine — Gemcitabine 800 mg/m2 in 250 mL of normal saline, given as fixed dose-rate (, 10 mg/m2/min) infusion, day 1; After the administration of gemcitabine, the infusion line should be flushed with 20 ml of normal saline and then 50 ml of 5% glucose solution before the administration of oxaliplatin. in SLOG arm.
  Gemcitabine 1000 mg/m2 in 100 mL of normal saline, IV drip for 30 mins on D1 and D8 ，in GC arm
  Other Names: Gemmis
  Arms: SLOG regimen
Drug: Cisplatin — Cisplatin 25 mg/m2 in 250ml of normal saline, IV drip for 2 hours on D1 and D8
  Arms: GC regimen

SUMMARY:
To evaluate the following items in patients with locally advanced and metastatic biliary tract cancer receiving SLOG or GC treatment, Primary objective: 6-month progression-free survival rate

Secondary objectives:

Objective response rate Disease control rate (Objective response rate (ORR) + stable disease ≧ 12 weeks) Progression-free Survival Overall survival Safety profile Biomarker study

DETAILED DESCRIPTION:
To evaluate the following items in patients with locally advanced and metastatic biliary tract cancer receiving SLOG or GC treatment, Primary objective: 6-month progression-free survival rate Secondary objectives: Objective response rate、Disease control rate (Objective response rate (ORR) + stable disease ≧ 12 weeks)、Progression-free Survival 、Overall survival 、 Safety profile、Biomarker study This is a randomized, open-labeled, two-arm, multi-center, phase II clinical study.

Arm 1: SLOG regimen: every 14 days as one cycle S-1 35 mg/m2/b.i.d., day 1 - 7 (maximum dose: 120 mg/day) Leucovorin 30 mg/b.i.d., day 1-7; Oxaliplatin 85 mg/m2 in 250 mL of 5% Glucose, given as 2-hour intra- venous infusion, day 1; Gemcitabine 800 mg/m2 in 250 mL of normal saline, given as fixed dose-rate (FDR, 10 mg/m2/min) infusion, day 1; After the administration of gemcitabine, the infusion line should be flushed with 20 ml of normal saline and then 50 ml of 5% glucose solution before the administration of oxaliplatin.

Arm2: GC regimen: every 21 days as one cycle Gemcitabine 1000 mg/m2 in 100 mL of normal saline, IV drip for 30 mins on D1 and D8 Cisplatin 25 mg/m2 in 250ml of normal saline, IV drip for 2 hours on D1 and D8

Treatment will be stopped in case of progressive disease, unacceptable toxicity, patients' refusal or death.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed, advanced or metastatic biliary tract carcinoma (including intrahepatic bile duct, hilum bile duct, extrahepatic bile duct and gallbladder), except ampulla vater cancer or combined hepatocholangiocarcinoma.
* presence of at least one measurable tumor lesion which is defined as lesions that can be accurately measured in at least 1 dimension with longest diameter (LD) ≥20 mm using conventional techniques or ≥10 mm with spiral CT and MRI; measurable lymph nodes must be≥15 mm in the short axis.
* Patients must have no history of prior chemotherapy for Biliary Tract Cancer, except those delivered as adjuvant setting that completed at least 6 months before documentation of recurrence by imaging study.
* Patients with prior radiotherapy are eligible if the irradiated area does not involve the only source of measurable / evaluable disease.
* Patients' baseline Eastern Cooperative Oncology Group (ECOG)performance status must be less than or equal 1.
* Patients' life expectancy must be 12 weeks or greater.
* Patients' age must be more than or equal 20 years old.
* Patients must have adequate bone marrow function, defined as white blood cell (WBC) count ≥3,500/ul, absolute neutrophil count (ANC) 1,500/ul, and platelet count ≥100,000/ul.
* Patients must have adequate liver function and adequate renal function, defined as the following: serum alanine (ALT) 3 times upper normal limit, serum total bilirubin level less than or equal 2.0 mg/dL, and creatinine clearance rate (CCr) ≥ 60 mL/min ((based upon 24-hour urine collection or calculated by Cockcroft-Gault formula).
* Patients with biliary obstruction and adequate drainage procedures before enrollment are eligible.
* Patients must agree to have indwelling venous catheter implanted.
* Women or men of reproductive potential should agree to use an effective contraceptive method.
* All patients must be informed of the investigational nature of this study and must sign and give written informed consent.

Exclusion Criteria:

* Patients who have major abdominal surgery, radiotherapy or other investigating agents within 4 weeks are not eligible. Patients who have palliative radiotherapy for bony metastasis will be eligible 2 weeks after the completion of radiotherapy.
* Patients with central nervous system metastasis
* Patients with active infection
* Pregnant or breast-nursing women
* Patients with active cardiopulmonary disease or history of ischemic heart disease
* Patients who have peripheral neuropathy > Grade I of any etiology, presence of grade 2 or above ascites or pleural effusion, or ≥ grade 2 of diarrhea.
* Patients who have serious concomitant systemic disorders incompatible with the study, i.e. poorly controlled diabetes mellitus, auto-immune disorders, cirrhosis of the liver, and the rest will be at the discretion of in-charged investigator.
* Patients who have other prior or concurrent malignancy except for adequately treated in situ carcinoma of cervix or adequately treated basal cell carcinoma of skin, or any malignancy remains disease-free for 3 or more years after initial curative treatment
* Patients who are under biologic treatment for their malignancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2018-04-19 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
6-month progression-free survival rate | From date of registration to the date of disease progression or date of death from any cause, whichever came first, assessed up to 26 weeks .
  Tumor response will be evaluated by Response Evaluation Criteria in Solid Tumors (RECIST)Guidelines version 1.1.

SECONDARY OUTCOMES:
tumor response | From date of registration to the date of disease progression or date of death from any cause, whichever came first, assessed up to 26 weeks .
  Efficacy evaluations: objective tumor response according to RECIST 1.1
Overall survival | Overall survival will be assessed. From date of registration until the date of death, assessed up to 60 months.
  Overall survival: defined as the time from the date of first study treatment to the date of patient death, due to any cause, or to the last date the patient was known to be alive. The primary analysis population for the overall survival will be per-protocol population. The endpoint will also be analyzed in the intent-to-treat population. Kaplan-Meier estimates will be calculated for the overall survival.
Disease control rate (Objective response rate (ORR) + stable disease ≧ 12 weeks) | From date of registration to the date of disease progression or date of death from any cause, whichever came first, assessed up to 26 weeks .
  Efficacy evaluations: objective tumor response according to RECIST 1.1
Safety profile | From date of registration to the date of disease progression or date of death from any cause, whichever came first, assessed up to 26 weeks .
  Adverse events (AEs) will be evaluated according to the National Cancer Institute's Common Terminology Criteria for Adverse Events version 4 (CTCAE v4).All required pre-treatment and interim data should be available and the physician must have made a designation as to response if a re-evaluation has been performed and the grade of toxicity if any has occurred。
Biomarker study | From date of registration to the date of disease progression or date of death from any cause or date of unacceptable toxicity or date of patient's refusal , whichever came first, assessed up to 26 weeks .
  evaluated for biomarkers, including inflammatory cytokine (TGF-β, hepatocyte growth factor (HGF), interleukin (IL)-6, IL-8, IL-1, CXCL-1, Chemokine (C-X-C motif) ligand 3(CXCL-3), and stromal-derived factor (SDF)...etc). Tumor DNA will be extracted from formalin-fixed paraffin-embedded(FFPE) slides for p53, CDKN2A and AT-rich interactive domain-containing protein 1A (ARID1A) mutation which were reported to be correlated with chemotherapy resistance

CONTACTS AND LOCATIONS:
Overall Officials: Li-Tzong Cheng, PHD, Study Chair — National Health Research Institute, Cancer Research
Locations (1):
- Taiwan Cooperative Oncology Group, National Health Research Institutes, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No